CLINICAL TRIAL: NCT05832099
Title: Cognition-preserving Brain Irradiation for Treating Patients With Intracranial Meningioma in the Era of Modern Radiotherapeutic Techniques Including Proton Beam Therapy - a Prospective Study Focusing on Radiological Outcomes and Neurocognitive Endpoints
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202202092A3
Record Dates: First submitted 2023-03-15; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Meningioma
Keywords: Intracranial Meningioma; Radiation Therapy; Magnetic Resonance Image (MRI); Volumetric MRI; Functional MRI (fMRI); Radiological Outcomes; Hippocampus; Neurocognitive Functions (NCFs); Cognition-Preserving Brain Radiotherapy; Proton Beam Radiotherapy; Hippocampal Atrophy; Amygdala; Thalamus
MeSH Terms: conditions — Meningioma | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiation: Conformal focal-brain irradiation using modern radiotherapeutic techniques (i.e., conventionally fractionated VMAT, hypofractionated stereotactic radiotherapy, and proton beam therapy, etc)
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — The techniques of conformal focal-brain irradiation in the era of modern radiotherapy (i.e., conventionally fractionated VMAT, hypofractionated stereotactic radiotherapy, and proton beam therapy, etc)

SUMMARY:
【Background】For cranial-irradiation-naive patients with intracranial meningiomas at risk of local recurrence, the administration of conformal cranial radiotherapy can enhance tumor control in the current era of modern radiotherapeutic techniques. Life expectancy in patients with intracranial meningiomas, particularly non-malignant meningiomas (WHO grade I and II) is essentially similar to people of general population. However, RT-related neurocognitive function (NCF) sequelae are potentially and seriously a concern which should not be ignored. In terms of the natural course of cranial irradiation-induced NCF decline, it might vary considerably according to the specific domains which are selected to be measured. Early neurocognitive decline principally involves impairments of episodic memory, which is significantly associated with functions of the hippocampus. Additionally, the extent of changes in hippocampal volume after local irradiation may be associated with the hippocampal dosimetry. This study thus aims to investigate the potential cause-effect relationship between the hippocampal dosimetry and radiological outcomes represented by the volumetric changes regarding the contralateral hippocampus; furthermore, the correlation between radiological outcomes and neurocognitive endpoints will be examined and clarified.

【Methods】Patients with cranial-RT-naive intracranial meningiomas may be eligible and therefore enrolled in this prospective study addressing both radiological outcomes and neurocognitive endpoints. All eligible and recruited patients should receive baseline volumetric brain MRI examination and baseline neurobehavioral assessment. Subsequently, conformal cranial irradiation in the era of modern radiotherapeutic techniques (including hypofractionated stereotactic radiotherapy, proton beam therapy volumetric modulated arc therapy) will be utilized in order to reduce the dose irradiating the contralateral hippocampus and other relevant organs at risk. The prescribed dose schemes for treating patients with intracranial meningioma depend on the decision of the radiation oncologist in charge and follow the treatment guidelines at our cancer center. Accordingly, a battery of neurocognitive measures, which includes 9 standardized neuropsychological tests categorized into 5 NCF domains (e.g., executive functions, verbal & non-verbal memory, working memory, psychomotor speed, and amygdala-related emotion recognition), is used to evaluate neurocognitive performances longitudinally for our registered patients. There will be two co-primary outcome measures in the current study. The main primary outcome will be the correlation between the mean hippocampal dose and the extent of change in hippocampal volume at 6 months after the course of cranial RT. The other primary endpoint will be 6-month cognitive-deterioration-free survival.

【Expected Results】This prospective observational cohort study aims to explore and investigate the cause-effect relationship between the hippocampal dosimetry (i.e., mean dose irradiating the hippocampus, particularly the one contralateral to the lateralization of intracranial meningioma) and the extent of hippocampal atrophy signifying one of the measures regarding radiological outcomes. Simultaneously, predefined standardized neurocognitive outcome measures such as hippocampus-related memory functions and amygdala-related emotion recognition will be obtained prospectively and longitudinally in order to examine whether any meaningfully significant correlation exists between the above radiological outcome measures and neurocognitive endpoints. The mutual associations among hippocampal dosimetry, radiological outcomes including the MRI-delineated hippocampal volume, and neurocognitive endpoints including hippocampus-related verbal/non-verbal memory functions will be examined thoroughly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically or pathologically-confirmed intracranial non-malignant meningiomas who are at least 18 years old, referred for arranging conformal radiotherapy
* A Fair/good performance status superior to Eastern Cooperative Group (ECOG) of 2 or an acceptable performance status of Karnofsky Score (KPS) at least 70

Exclusion Criteria:

* History of prior radiotherapy delivered to brain/head region for any reason, including stereotactic radiosurgery
* Patients with malignant meningiomas diagnosed pathologically (WHO grade III)
* Patients with presumed clinical target volume (CTV) encompassing bilateral peri-hippocampal regions within 5 mm away from the adjacent periphery of the hippocampus
* Patients whose quality of volumetric MRI fails to meet the minimal requirements for physicians to delineate the hippocampal contouring (i.e., slice thickness > 2mm)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically or pathologically-confirmed intracranial non-malignant meningiomas referred for arranging conformal focal-brain irradiation using modern radiotherapeutic techniques including volumetric modulated arc therapy (VMAT), hypofractionated stereotactic radiotherapy (SRT), and proton beam therapy.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes in the volumes of organs at risk including the hippocampus | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Longitudinal changes in the volumes (cc) of the left hippocampus, right hippocampus, left amygdala, right amygdala, left thalamus, right thalamus, and so on based on volumetric MR imaging examinations

SECONDARY OUTCOMES:
Change in verbal memory function | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Change in verbal memory function related to left hippocampus from baseline to 4 months after cognition-preserving cranial RT
Change in non-verbal memory learning | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Change in non-verbal memory learning associated with right hippocampus from baseline to 4 months after cognition-preserving brain RT
Change in executive function | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Change in executive function related to hippocampus from baseline to 4 months after cognition-preserving cranial RT.
  Concerning the domain of executive functions generally dominated by the frontal lobes, the Modified Card Sorting Test is employed to assess both conceptual formation and mental shifting which have been documented to be the major components of executive functions.
Change in emotion memory task | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Change in emotion memory tasks associated with the amygdala from baseline to 4 months after cognition-reserving cranial irradiation.
  For evaluate and quantify the cognitive function of amygdala, the NCF test tailored to the emotional recognition task will be used and patients' performances will be assessed using the commercialized and computerized test included in Cambridge Cognition® package.
Change in working memory | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Change in working memory related to hippocampus from baseline to 4 months after cognition-preserving cranial RT.
  Working memory includes executive functions and psychomotor speed.
  * The neurocognitive outcome of verbal working memory was determined by the Digit Span Subtest (DS) and Spatial Span (SSP) of the Wechsler Adult Intelligence Scale- 3rd edition (WAIS-III®).
  * In order to indicate patients' performance on the psychomotor speed, we make use of Psychomotor Speed Index (PSI), which is derived from the composite score of Digit Symbol Coding Subtest (DSS) and Symbol Searching Subtest (SS) of the WAIS-III®.
Longitudinal changes in the imaging biomarkers | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Longitudinal changes in the imaging biomarkers from DTI imaging
Longitudinal changes in the fractional anisotropy | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Longitudinal changes in the fractional anisotropy (FA, unitless index between 0 and 1) from DTI imaging
Trajectories in the imaging biomarker | baseline (pre-RT), 4 months, 8-10 months (optional), 12 months, 18 months, 24 months
  Trajectories in the imaging biomarker, mean diffusivity (MD, mm squared/second) based on DTI imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan